CLINICAL TRIAL: NCT00947843
Title: Assessment of the Efficacy and Tolerability of Clopidogrel Resinate and Clopidogrel Bisulfate in Patients With Coronary Heart Disease (CHD) or CHD Equivalents : A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Tolerability of Clopidogrel Resinate and Clopidogrel Bisulfate in Patients With Coronary Heart Disease (CHD) or CHD Equivalents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: CKD Pharmaceutical Limited (Unknown)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Principal investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KOPRE-DM/CAD
Record Dates: First submitted 2009-07-25; First posted 2009-07-28 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Heart Disease
Keywords: CHD; CHD equivalents
MeSH Terms: conditions — Coronary Disease | interventions — Aspirin; clopidogrel resinate; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- aspirin+placebo (Placebo Comparator): aspirin protect (Bayer) 100mg + placebo clopidogrel 75mg for 1mo
  Interventions: Drug: aspirin + placebo
- aspirin+pregrel (Active Comparator): pregrel is a generic brand name of clopidogrel
  Interventions: Drug: aspirin + pregrel (Clopidogrel resinate)
- Aspirin+Plavix (Active Comparator): plavix is a original brand name of clopidogrel
  Interventions: Drug: aspirin + plavix (Clopidogrel bisulfate)

INTERVENTIONS:
Drug: aspirin + pregrel (Clopidogrel resinate)
  Other Names: Aspirin: Aspirin Protect (Bayer) 100mg; Pregrel: Clopidogrel resinate (CKD Pharmaceutical) 75mg
  Arms: aspirin+pregrel
Drug: aspirin + placebo
  Arms: aspirin+placebo
Drug: aspirin + plavix (Clopidogrel bisulfate)
  Other Names: aspirin : Aspirin Protect (Bayer) 100mg; plavix : Clopidogrel bisulfate (Sanofi-Aventis) 75mg
  Arms: Aspirin+Plavix

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability between clopidogrel resinate and clopidogrel bisulfate in patients with coronary heart disease (CHD) or CHD equivalents.

ELIGIBILITY:
Inclusion Criteria:

* Korean men and women aged 20 to 85 years with coronary heart disease (CHD) or CHD equivalent patients
* Atherosclerotic plaques in coronary computed tomography (CT) or angiography or
* History of PCI or coronary artery bypass graft surgery (CABG) > one year or
* Diabetes mellitus (including type I and type II) or
* Confirmed carotid atherosclerotic plaque with sonography, CT or angiography or
* History of peripheral artery disease or
* History of cerebrovascular disease

Exclusion Criteria:

* Patients who had history of PCI within one year
* Patients who used concomitant anticoagulants
* Patients who had hypersensitivity to aspirin or clopidogrel, serious bleeding tendency, history of intracranial hemorrhage, sign of active bleeding, uncontrolled hypertension
* Chronic alcoholism or drug addiction
* Women who were pregnant or breastfeeding or who were not using an effective method of contraception
* The use of glycoprotein IIb/IIIa inhibitor, daily NSAIDs, lipid lowering agent (except atorvastatin), or substances with possible interactions with the study drug

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The percentage of P2Y12 receptor inhibition assessed by Ultegra rapid platelet function analyzer, (Baseline platelet reaction unit (PRU)- posttreatment PRU)/Baseline PRU * 100 (%)) | 1 month

SECONDARY OUTCOMES:
Adverse events after study medication | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bae Seung, MD, PhD, Study Director — Seoul St. Mary's Hospital; Chung-Hwan Gwak, MD, PhD, Study Director — Gyeongsang National University Hospital; Kwon-Sam Kim, MD,PhD, Study Director — Kyung Hee University Hospital; Soon-Jun Hong, MD,PhD, Study Director — Korea University Anam Hospital; Tae-Ho Park, MD,PhD, Study Director — Dong-A medical center; Sang-Hyun Kim, MD,PhD, Study Director — Seoul Metropolitan Boramae Hospital; Seung-Jea Tahk, MD,PhD, Study Director — Ajou University Medical Center; Seung-Jae Joo, MD,PhD, Study Director — Jeju National University Hospital; Young-Jin Choi, MD,PhD, Study Director — Hallym University Medical Center

REFERENCES:
- [Derived] Suh JW, Seung KB, Gwak CH, Kim KS, Hong SJ, Park TH, Kim SH, Choi YJ, Joo SJ, Tahk SJ, Kim HS. Comparison of antiplatelet effect and tolerability of clopidogrel resinate with clopidogrel bisulfate in patients with coronary heart disease (CHD) or CHD-equivalent risks: a phase IV, prospective, double-dummy, parallel-group, 4-week noninferiority trial. Clin Ther. 2011 Aug;33(8):1057-68. doi: 10.1016/j.clinthera.2011.07.001. Epub 2011 Aug 4. PMID 21816478